CLINICAL TRIAL: NCT00141154
Title: A Randomized, Multicenter, Active And Placebo Controlled Parallel Group Study To Evaluate The Efficacy And Safety Of Celecoxib (Ym177) 200 Bid Compared To Loxoprofen 60 Mg Tid In Patients With Low Back Pain
Brief Title: Comparison Of Celecoxib 200 Mg Bid, Loxoprofen Sodium 60 Mg Tid And Placebo In Low Back Pain In Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191174
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Celecoxib; loxoprofen

INTERVENTIONS:
Drug: Celecoxib
Drug: Placebo
Drug: Loxoprofen

SUMMARY:
To verify the superiority of celecoxib (YM177) 200 mg bid to placebo in treatment of patients with low back pain as well as non-inferiority to loxoprofen sodium 60 mg tid.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have the major site of the low back pain at the 12th thoracic vertebra or lower
* Patients who have had low back pain for at least two weeks

Exclusion Criteria:

* Patients who have a previous history or complication of rheumatoid arthritis, spondylarthrosis with negative serum reaction (ankylosing spondylarthritis, psoriatic arthritis), metastasis of tumor, Paget's disease, fibromyalgia, tumor or infection of spinal cord or intervertebral disc, or any other disease which can cause systemic pain

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1234 (Actual)
Dates: Start 2004-10

PRIMARY OUTCOMES:
Patient's pain assessment (VAS: Visual Analogue Scale)

SECONDARY OUTCOMES:
Patient's global assessment (VAS), Physician's global assessment (VAS), Roland Morris Disability Questionnaire (RDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- Japan (36):
  - Pfizer Investigational Site, Funabashi, Chiba
  - Pfizer Investigational Site, Funabashi-shi, Chiba
  - Pfizer Investigational Site, Matsudo-shi, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Chitose, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Katougun, Hyōgo
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Nishinomiya, Hyōgo
  - Pfizer Investigational Site, Sagamihara-shi, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Hatogaya-shi, Saitama
  - Pfizer Investigational Site, Kumagaya-shi, Saitama
  - Pfizer Investigational Site, Kumagayashi, Saitama
  - Pfizer Investigational Site, Minamisaitama-gun, Saitama
  - Pfizer Investigational Site, Saitama-shi, Saitama
  - Pfizer Investigational Site, Tokorozawa, Saitama
  - Pfizer Investigational Site, Adachi-Ku, Tokyo
  - Pfizer Investigational Site, Bunkyou-ku, Tokyo
  - Pfizer Investigational Site, Edogawa-ku, Tokyo
  - Pfizer Investigational Site, Itabashi-ku, Tokyo
  - Pfizer Investigational Site, Koito-ku, Tokyo
  - Pfizer Investigational Site, Meguro-Ku, Tokyo
  - Pfizer Investigational Site, Nakano-ku, Tokyo
  - Pfizer Investigational Site, Nerima-ku, Tokyo
  - Pfizer Investigational Site, Ōta-ku, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shibuya-ku, Tokyo
  - Pfizer Investigational Site, Shinagawa-ku, Tokyo
  - Pfizer Investigational Site, Shinjyuku-ku, Tokyo
  - Pfizer Investigational Site, Suginami-ku, Tokyo
  - Pfizer Investigational Site, Sumida-ku, Tokyo
  - Pfizer Investigational Site, Toyoshima-ku, Tokyo
  - Pfizer Investigational Site, Chiba
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191174&StudyName=Comparison+Of+Celecoxib+200+Mg+Bid%2C+Loxoprofen+Sodium+60+Mg+Tid+And+Placebo+In+Low+Back+Pain+In+Japan